CLINICAL TRIAL: NCT00430391
Title: Comparison of Video Consent and Routine Consent for Research
Brief Title: Comparison of Video Consent Versus Routine Consent for Participation in Research Studies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Dilip V. Jeste, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: R01MH067902 (NIH); R01MH067902 (NIH)
Record Dates: First submitted 2007-01-31; First posted 2007-02-01 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2011-01

CONDITIONS: Schizophrenia
Keywords: DVD; Multi-media; Schizophrenia; Normal Comparison; Consent procedures
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- DVD patient high risk (Experimental): Patients with a diagnosis of schizophrenia/schizoaffective disorder randomized to the DVD, high risk version
  Interventions: Other: DVD Consent
- DVD patient low risk (Experimental): Patient with a diagnosis of schizophrenia/schizoaffective disorder randomized to DVD consent, low risk version
  Interventions: Other: DVD Consent
- DVD normal high risk (Experimental): Participants with no psychiatric diagnosis randomized to DVD consent, high risk version
  Interventions: Other: DVD Consent
- DVD normal low risk (Experimental): Participants with no psychiatric diagnosis randomized to DVD consent, low risk version
  Interventions: Other: DVD Consent
- Routine control high risk (Experimental): Participants with no psychiatric diagnosis randomized to routine consent, high risk version
  Interventions: Other: Routine Control
- Routine control low risk (Experimental): Participants with no psychiatric diagnosis randomized to routine consent, low risk version
  Interventions: Other: Routine Control
- Routine patient low risk (Experimental): Participants with schizophrenia/schizoaffective disorder randomized to routine consent, low risk version
  Interventions: Other: Routine Control
- Routine patient high risk (Experimental): Participants with schizophrenia/schizoaffective disorder randomized to routine consent, high risk version
  Interventions: Other: DVD Consent; Other: Routine Control

INTERVENTIONS:
Other: DVD Consent — Participants are randomized to DVD enhanced consent that is either high risk or low risk.
  Arms: DVD normal high risk; DVD normal low risk; DVD patient high risk; DVD patient low risk; Routine patient high risk
Other: Routine Control — Participants are assigned to the routine, standard consent.
  Arms: Routine control high risk; Routine control low risk; Routine patient high risk; Routine patient low risk

SUMMARY:
The purpose of this study is to examine a novel technique for improving the informed consent process for participation in research by the older psychiatric population.

DETAILED DESCRIPTION:
This study will test a new method of delivering informed consent procedures to people with schizophrenia. The study has two aims. First, it will examine the impact of a multimedia DVD-based informed consent process on the ability of participants to make decisions regarding participation in research, both after the initial presentation of information and after 1 month. Second, it will examine the association between participant personal characteristics and the benefit derived from the DVD-based informed consent process.

Participants with schizophrenia and a normal comparison group will participate in either a routinely used informed consent procedure or an enhanced, DVD-based informed consent procedure. The outcome measure, comprehension of the consent materials, including understanding of the risks and benefits of participating in the study, will be assessed in each group. It is expected that the normal control group will reach the requisite level of comprehension faster than the schizophrenia group.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of schizophrenia or no current or past major neuropsychiatric disorder (normal subjects)
* Fluency in English
* Written informed consent

Exclusion Criteria:

* Known or suspected dementia

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 382 (Actual)
Dates: Start 2003-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Comprehension of the consent materials, including understanding of the risks and benefits of participating in the study | Measured at 1-month follow-up

SECONDARY OUTCOMES:
Association of subject characteristics with the degree of benefit derived from the DVD-based consent over routine consent procedure | Measured at 1-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Dilip V. Jeste, MD, Principal Investigator — UCSD
Locations (1):
- University of California, San Diego, San Diego, California, United States